CLINICAL TRIAL: NCT01543880
Title: Non-interventional Study of Safety and Efficacy of Long-term Somatropin Treatment in Adults
Brief Title: Safety and Efficacy of Long-term Somatropin Treatment in Adults
Acronym: NordiWIN
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: GH-1931
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Growth Hormone Disorder; Adult Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Users of somatropin
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — Prescribed at the discretion of the treating physician according to product labelling

SUMMARY:
This study is conducted in Europe. The aim of the study is to evaluate safety and efficacy in adults treated with somatropin (Norditropin®).

ELIGIBILITY:
Inclusion Criteria:

* In need of somatropin or current user

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults in need of somatropin or current users
Sampling Method: Probability Sample
Enrollment: 752 (Actual)
Dates: Start 2003-07; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | Up to 10 years

SECONDARY OUTCOMES:
BMI (Body Mass Index) | Up to 10 years
HbA1c change | Up to 10 years
IGF-I (Insulin-Like Growth Factor I) | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Mainz, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com